CLINICAL TRIAL: NCT07355764
Title: SHR-1811 Combined With Bevacizumab as Second-line Treatment in Patients Metastatic CRC
Brief Title: MA-CRC-II-016 SHR-1811
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xicheng Wang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: K8750; K8750 (Registry Identifier: Peking union medical college hospital ethics committee)
Record Dates: First submitted 2025-12-17; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: mCRC; HER2; Targeted Therapy; Antibody-drug Conjugates
Keywords: SHR-1811; mCRC; second-line
MeSH Terms: interventions — Bevacizumab; Drug Therapy

STUDY DESIGN:
Intervention Model Description: SHR-A1811 combined with bevacizumab; chemotherapy combined with bevacizumab
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1811 combined with bevacizumab (Active Comparator): SHR-A1811 with bevacizumab
  Interventions: Drug: SHR-A1811 & Bevacizumab injection
- Chemotherapeutic Combinations (Active Comparator): chemotherapy with bevacizumab
  Interventions: Drug: Chemotherapeutic Combinations

INTERVENTIONS:
Drug: SHR-A1811 & Bevacizumab injection — HER2 ADC
  Other Names: bevacizumab; chemotherapy
  Arms: SHR-A1811 combined with bevacizumab
Drug: Chemotherapeutic Combinations — FOLFIRI+BEV
  Arms: Chemotherapeutic Combinations

SUMMARY:
A randomized, controlled, multicenter clinical study of SHR-A1811 combined with bevacizumab for the second-line treatment of metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

-Provide a written informed consent form to voluntarily participate in this study.

Male or female subjects aged 18-75 years.

* Patients with histologically or cytologically confirmed recurrent or metastatic colorectal adenocarcinoma that is not amenable to curative resection.
* Patients who have experienced disease progression following first-line standard therapy with oxaliplatin combined with fluoropyrimidine-based drugs.
* Patients with disease progression within 12 months after completion of neoadjuvant or adjuvant therapy are eligible for inclusion.
* Patients who have previously received irinotecan as part of first-line therapy may be included if investigators from the leading center determine through discussion that the patient is likely to benefit from treatment in the control group.
* HER2 expression status: Includes patients with HER2 overexpression (IHC 3+ / IHC 2+ with FISH positivity) or HER2 low-to-moderate expression (IHC 2+ with FISH negativity or IHC 1+).
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1.
* Ability to provide a report documenting RAS/BRAF gene status.
* Expected survival time of at least 6 months.
* Presence of radiologically assessed measurable lesions at baseline (per RECIST 1.1 criteria). Measurable lesions should not have received prior local therapy such as radiotherapy. Lesions located within previously irradiated areas may be selected as target lesions if disease progression in these lesions is confirmed.
* Adequate function of major organs, meeting the following requirements (administration of blood components or cell growth factors for corrective treatment is not allowed within 14 days prior to the first dose of study medication):
* Absolute Neutrophil Count (ANC) ≥ 1.5 × 10⁹/L Platelet count ≥ 100 × 10⁹/L Hemoglobin ≥ 90 g/L Serum albumin ≥ 30 g/L Total bilirubin ≤ 1.5 × Upper Limit of Normal (ULN) Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 2.5 × ULN; for patients with liver metastases, ALT and AST ≤ 5 × ULN Serum creatinine ≤ 1.5 × ULN or creatinine clearance rate > 60 mL/min (calculated by the Cockcroft-Gault formula) Activated Partial Thromboplastin Time (APTT) and International Normalized Ratio (INR) ≤ 1.5 × ULN. Patients receiving stable-dose anticoagulant therapy (e.g., low-molecular-weight heparin or warfarin) with INR within the expected therapeutic range for anticoagulants are eligible for screening.
* For female subjects of childbearing potential:

A negative serum pregnancy test result is required within 3 days prior to the first dose, and the subject must not be breastfeeding.

Must agree to use effective contraceptive measures during the study period and for at least 7 months after the last dose of SHR-A1811, or for at least 6 months after the last dose of other study medications.

-For male subjects whose partners are of childbearing potential: The subject must have undergone surgical sterilization, or agree to use effective contraceptive measures during the study period and for at least 7 months after the last dose of SHR-A1811, or for at least 6 months after the last dose of other study medications.

Sperm donation is prohibited during the study period.

Exclusion Criteria:

* Toxicities from prior anti-tumor therapies have not resolved to ≤ Grade 1 per the CTCAE v5.0 criteria (except for toxicities deemed to pose no safety risk by the investigator, e.g., alopecia) or to the levels specified in the inclusion/exclusion criteria.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with a history of treated brain metastases may be enrolled provided that their brain metastases are stable, and they have not received steroid therapy for brain metastases for at least 28 days prior to study initiation. This exception does not apply to carcinomatous meningitis, as patients with carcinomatous meningitis are excluded regardless of clinical stability.
* Known microsatellite instability-high (MSI-H) status confirmed by genetic testing or deficient mismatch repair (dMMR) status confirmed by immunohistochemistry.
* A history of hypersensitivity to monoclonal antibodies, the formulation components of SHR-A1811, or anti-angiogenic agents.
* Prior treatment with HER2-targeted antibody-drug conjugates (ADCs).
* Major surgery, open biopsy, or severe trauma within 28 days prior to the first study drug administration.
* Patients with any severe and/or uncontrolled diseases, including:

Patients with inadequately controlled hypertension; Myocardial ischemia or myocardial infarction of Grade ≥1, cardiac arrhythmias (including QT interval ≥ 480 ms), or cardiac insufficiency of Grade ≥1; Active or uncontrolled severe infections; Hepatic diseases such as decompensated liver disease, active hepatitis B (HBV-DNA ≥ 10⁴ copies/mL or 2000 IU/mL) or active hepatitis C (positive for hepatitis C antibody with HCV-RNA level above the lower limit of quantification of the assay); Subjects with urine protein ≥ ++ on routine urinalysis and confirmed 24-hour urine protein quantification > 1.0 g.

* Clinically significant bleeding symptoms or confirmed bleeding diathesis (e.g., gastrointestinal bleeding, hemorrhagic gastric ulcer, or vasculitis) within 3 months prior to the first study drug administration.
* Arterial/venous thrombotic events (e.g., cerebrovascular accident including transient ischemic attack, cerebral hemorrhage, cerebral infarction; deep vein thrombosis; pulmonary embolism) within 6 months prior to the first study drug administration. Subjects with superficial venous thrombosis may be enrolled at the investigator's discretion.
* Presence of another concurrent progressive malignancy requiring active treatment, with the exception of non-melanoma skin cancer and carcinoma in situ of the cervix that have undergone potential curative treatment.
* Any other factors judged by the investigator that may force the subject to discontinue the study prematurely, including severe concurrent illnesses (including mental illnesses) requiring concomitant treatment, severely abnormal laboratory test results, family or social factors that may affect subject safety or the collection of trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
ORR | The end of cycle 2 (each cycle is 21 days) for SHR-A1811+BEV group and the end of cycle 3 (each cycle is 14 days) for FOLFIRI+BEV group
  objective response rate

SECONDARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  progression free survival
OS | From data of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  overall survival